CLINICAL TRIAL: NCT07207096
Title: Observational Case Series of Patients With Parkinson's Disease (PD) Attending a Complementary Medicine Neuro-degenerative Disease (NDD) Clinic.
Status: Recruiting | Type: Observational
Sponsor: St. Mary's University, Twickenham (Other)
Collaborators: Faculty of Homeopathy (Unknown); Homeopathy UK (Unknown)
Responsible Party: Principal Investigator, Philippa Fibert, associate lecturer, St. Mary's University, Twickenham
Other Study IDs: SMU_ETHICS_2024_25_1128
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: homeopathy; herbalism; hypnosis; healing; complementary medicine; lifestyle; self-help; mindfulness; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Complementary Therapies; Homeopathy; Hypnosis; Mindfulness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: complementary medicine — Complementary therapies provided include homeopathy, herbalism, hypnosis, and healing. Patients may also be provided with self-help advice for lifestyle changes, mindfulness or meditation techniques, and dietary advice, as indicated for complementary therapy management of their condition.
  Other Names: homeopathy; herbalism; hypnosis; healing; self-help and lifestyle advice; mindfulness

SUMMARY:
When the charity Homeopathy UK launched a new London based charitable clinic for Neurodegenerative Diseases (NDD), including Parkinson's Disease (PD), it was considered important to document patient's experiences of a high-quality complementary medicine clinic, to enable a greater understanding of the role of complementary medicine for PD.

Routine clinical data, including a couple of questionnaires, is collected from consecutive patients with PD seen in the NDD clinic. Treatments provided are complementary to patients' usual medical treatment, and include homeopathy, herbalism, hypnosis, and healing. Patients may also be provided with self-help advice for lifestyle changes, mindfulness or meditation techniques, and dietary advice, as indicated for complementary therapy management of their condition. Consultations take place approximately every 3 months and patients complete questionnaires at the time of each consultation.

DETAILED DESCRIPTION:
Clinical research documenting the effectiveness of complementary medicine for PD is long overdue. Despite high rates of utilization, data on efficacy is generally limited, restricting physicians in providing guidance to interested patients (Bega, 2014).

When the charity Homeopathy UK launched a new London based charitable clinic specifically for NDD, including Parkinson's Disease, it was considered important to document patient's experiences of a high-quality complementary medicine clinic, to enable a greater understanding of the role of complementary medicine for PD.

This is an observational case series with no deviation from routine clinical practice. Routine clinical data is collected from consecutive PD patients seen in the NDD clinic. Patients complete questionnaires regardless of whether they take part in the research. Consultations take place approximately every 3 months (time between appointments may be reduced to 1 month for those patients needing more frequent management, or extended to 6 months for those who require less management). For those patients who are unable to travel, e.g. due to neurological disability and/or long distance away, the 1.5 hour appointment is provided as a remote clinic link using a secure zoom platform.

Treatments provided are complementary, i.e. provided alongside patients' usual medical treatment. Complementary therapies provided include homeopathy, herbalism, hypnosis, and healing. Patients may also be provided with self-help advice for lifestyle changes, mindfulness or meditation techniques, and dietary advice, as indicated for complementary therapy management of their condition.

Two validated outcome measures are used at each clinic visit. Both measures are used both for clinical assessment and the Observational Case Series.

* The MDS-sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) which has four parts. The majority of the MDS-UPDRS is completed by the clinic doctor, however Part IB is completed independently by the patient with or without the aid of the caregiver.
* Measure Your Own Medical Outcome Profile (MYMOP) is a patient generated outcome measure consisting of 4 self-chosen items measured using a likert type scale of 0 (as good as it could be) to 6 (as bad as it could be): two symptoms considered most bothersome, an activity which the condition limits participation in, and wellbeing.

It is a validated, personalized measure allowing patients to select their key concerns, and considered appropriate to capture the non-specific effects of complementary medicine.

We aim to collect routine data from 100+ consecutive PD patients. Patients are recruited to the observational study after they have booked an appointment for complementary therapy in the NDD clinic, and report a diagnosis of PD. Patients are informed of the study then and also during their initial clinic appointment. They are informed there is no compulsion to enrol into the study, and they can continue being assessed and treated at the clinic even if they remain outside the study, and that there is no difference in the standard of their treatment.

Bega, D., Gonzalez-Latapi, P., Zadikoff, C., & Simuni, T. (2014). A review of the clinical evidence for complementary and alternative therapies in Parkinson's disease. Current treatment options in neurology, 16, 1-19.

ELIGIBILITY:
Inclusion Criteria: A diagnosis of Parkinson's Disease (self-reported), and Parkinsonism from any causes (patients may have co-existing other health conditions)

Exclusion Criteria: Patients requiring acute medical assessment and management, (as this is beyond the scope of this clinic service) Patients with any other NDD condition Patients without a diagnosis of PD/Parkinsonism. E.g. those at risk of PD such as through a family history (patients in this category may receive treatment at the clinic but are not included in the Observational Case series.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who book an appointment for complementary therapy in the NDD clinic, and report a diagnosis of PD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The MDS-sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At each consultation (approximately every 3 months)
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications).
  The majority of the MDS-UPDRS is completed by the clinic doctor. However Part IB is completed independently by the patient with or without the aid of the caregiver.
Measure Your Own Medical Outcome Profile (MYMOP) | At each consultation (approximately every 3 months)
  MYMOP is a patient generated outcome measure consisting of 4 self-chosen items measured using a likert type scale of 0 (as good as it could be) to 6 (as bad as it could be): two symptoms considered most bothersome, an activity which the condition limits participation in, and wellbeing.
  It is a validated, personalized measure allowing patients to select their key concerns, and considered appropriate to capture the non-specific effects of complementary medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- Feldy Community Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be kept for a period of ten years on the St Mary's University Open Research Archive, which is a condition of St Mary's University